CLINICAL TRIAL: NCT01290406
Title: A Phase II, Single-arm Study of Orally Administered BEZ235 as Second-line Therapy in Patients With Advanced or Metastatic Endometrial Carcinoma
Brief Title: BEZ235 Trial in Patients With Advanced Endometrial Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBEZ235C2201; 2010-024396-12 (EudraCT Number); EudraCT 2010-024396-12 (Registry Identifier: EudraCT)
Record Dates: First submitted 2011-02-03; First posted 2011-02-07 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Endometrial Cancer
Keywords: Endometrial cancer,; uterine cancer,; PI3K,; mTOR,; targeted therapy
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Neoplasms | interventions — dactolisib

ARMS (1):
- BEZ235 (Experimental)
  Interventions: Drug: BEZ235

INTERVENTIONS:
Drug: BEZ235

SUMMARY:
This is an open label and single arm study to investigate the safety and efficacy of BEZ235 in adult women with endometrial carcinoma whose disease progressed (or recurred) while on or after first-line antineoplastic treatment for advanced endometrial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Female ≥ 18 years
* Histological confirmed diagnosis of advanced endometrial carcinoma with available tissue specimen, either archival tissue or fresh formalin fixed tumor biopsy
* Objective and radiologically confirmed progression of disease after prior first-line treatment
* Recovery (to grade ≤ 1) from all clinically significant toxicities related to prior therapies (except alopecia) with adequate bone marrow and organ functions
* At least one measurable lesion as per RECIST
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2

Exclusion Criteria:

* Previous treatment with PI3K and/or mammalian Target Of Rapamycin (mTOR) inhibitors
* More than one line of prior treatment for advanced or metastatic disease
* Active uncontrolled or symptomatic Central Nervous System (CNS) metastases
* Concurrent malignancy or malignancy in the last 3 years prior to start of study treatment
* Wide field radiotherapy ≤ 28 days or limited field radiation for palliation ≤ 14 days prior to enrollment in this study
* Active cardiac disease (e.g. Left Ventricular Ejection Fraction (LVEF) < 50%, Q-T interval corrected for heart rate (QTcF) > 480 msec on screening Electrocardiogram (ECG), unstable angina pectoris, ventricular, supraventricular or nodal arrhythmias)
* Inadequately controlled hypertension
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BEZ235
* Drugs with a known risk to induce Torsades de Pointes, moderate and strong inhibitors or inducers of CYP3A4, warfarin and coumadin analogues, Luteinizing Hormone-Releasing Hormone (LHRH) agonists
* Pregnant or nursing (lactating) woman

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2014-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
assess the efficacy of BEZ235 as measured by Overall Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) | every 8 weeks

SECONDARY OUTCOMES:
evaluate additional efficacy parameters (e.g. Disease Control Rate, Progression-Free Survival) | every 8 weeks
evaluate safety of BEZ235. Safety assessments will include vital signs, laboratory tests, and frequency of adverse events (non-serious and serious). | Treatment start until 30 days after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (59):
- United States (16):
  - St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - City of Hope Medical center, Duarte, California
  - Holy Cross Hospital, Silver Spring, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Morriswon Memorial Hospital, Morristown, New Jersey
  - Carolinas Healthcare Systems, Charlotte, North Carolina
  - Cancer Centers of North Carolina, Raleigh, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - GHS, Danville, Pennsylvania
  - Sarah Gautam Rau, Nashville, Tennessee
  - Texas Oncology, P.A., Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - STOH, San Antonio, Texas
  - Pacific Gynecology Specialists, Seattle, Washington
  - Cancer Care Northwest, Spokane, Washington
- Brazil (2):
  - Novartis Investigative Site, Rio de Janeiro
  - Novartis Investigative Site, São Paulo
- Canada (4):
  - Novartis Investigative Site, Hamilton
  - Novartis Investigative Site, Montreal
  - Novartis Investigative Site, Toronto
  - Novartis Investigative Site, Vancouver
- France (10):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, La Roche-sur-Yon
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Saint-Brieuc
  - Novartis Investigative Site, Toulouse
- Germany (7):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, München
- Italy (9):
  - Novartis Investigative Site, Aviano
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Brescia
  - Novartis Investigative Site, Capmobso
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Modena
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Roma
- Japan (3):
  - Novartis Investigative Site, Aichi
  - Novartis Investigative Site, Hyōgo
  - Novartis Investigative Site, Tokyo
- Poland (2):
  - Novartis Investigative Site, Środa Wielkopolska
  - Novartis Investigative Site, Warzawa
- Novartis Investigative Site, Saint Petersburg, Russia
- Novartis Investigative Site, Singapore, Singapore
- Spain (3):
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Oviedo
  - Novartis Investigative Site, Valencia
- Novartis Investigative Site, Istanbul, Turkey (Türkiye)